CLINICAL TRIAL: NCT01274910
Title: Effect of Fish Oil on Surgery Pain After Knee Replacement Patients: Randomized, Prospective, Double Blind, Placebo Control Trial
Acronym: EFOPaKR-01
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Pierre singer, Professor, MD, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5961
Record Dates: First submitted 2011-01-04; First posted 2011-01-12 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Fish Oil; Knee; Analgetics
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fish oil group (Active Comparator): Treatment Group.
  Interventions: Dietary Supplement: EPAX 6000 EE 1000mg (0.6 gr DHA+EPA)
- Control group (Placebo Comparator): Placebo group
  Interventions: Dietary Supplement: Capsules (Placebo)

INTERVENTIONS:
Dietary Supplement: EPAX 6000 EE 1000mg (0.6 gr DHA+EPA) — Patient will receive Fish Oil capsules (EPAX 6000 EE) .
  Treatment: 5 capsules per day
  Other Names: Caps.Omeguard Triomar 1000 mg SGC
  Arms: Fish oil group
Dietary Supplement: Capsules (Placebo) — Patient will receive capsules which not contain fish oil.
  Treatment: 5 capsules per day
  Arms: Control group

SUMMARY:
This is a single-center, prospective, randomized, double blind, placebo control study. The aim of this study is to assess the effect of fish oil capsules on pain intensity and postoperative analgesics consumption in patients after knee replacement surgery.

The study population will be adult are referred for knee replacement surgery due to osteoarthritis of the knee.

DETAILED DESCRIPTION:
Primary outcome:

Post surgical pain level and analgesics use

Secondary outcomes:

1. Pain levels and analgesic use at six weeks and 3 months after surgery
2. ω3 incorporation into blood cell membranes(RBC)
3. Stress and inflammation markers
4. Rates of postoperative complications

Study Procedure :

Enrolled patient will be randomly divided into a control group and intеrvention group during preoperative clinic visit. Each patient will receive total 150 capsules (5 capsules per day) accordingly to randomized group.

Patients in treatment group will receive Fish Oil capsules. Patients in control group will receive placebo capsules.

ELIGIBILITY:
Inclusion Criteria:

Patients are referred for knee replacement surgery due to osteoarthritis of the knee

* Exclusion Criteria:

  * Use of steroids, NSAIDs two weeks before surgery, antidepression drugs, antiepileptic drugs, coumadin
  * Diabetic neuropathy
  * Herpes-zoster/ post-herpetic neuralgia
  * n-3 supplements use

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-12 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Pain Levels | 10 weeks
  Pain assessment of patients will be measured using visual analog scale (VAS) score.
Analgetics use | 10 weeks
  All analgetics drugs used by patient will be noted

SECONDARY OUTCOMES:
Inflammatory Markers | Day 1
  Blood test. Concentration of circulated inflammatory markers (TNF-α,IL-1,IL-6).
Fatty Acids Composition | Day 1
  ω3 incorporation into blood cell membranes(RBC)
Cortisol | Day 1
  Cortisol levels in blood test.
ACTH | Day 1
  ACTH levels in blood test.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Singer, Professor, MD, Principal Investigator — ICU dep't, Rabin MC,Petah Tikva, Israel; Milana Grinev, RN, Study Coordinator, Study Director — ICU dep't, Rabin MC, Petah Tikva, Israel
Locations (1):
- Rabin Medical Center, Campus Beilinson, Petah Tikva, Petah Tikva, Israel